CLINICAL TRIAL: NCT01474980
Title: Retrospective Study :Describe the Changes of the Disease in Many Cases Likely to Aggravate.
Brief Title: Pregnancy Outcomes in Congenital Myasthenie Syndrome
Acronym: POCoMS
Status: Completed | Type: Observational
Sponsor: Institut de Myologie, France (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Laurent Servais, M.D., Laurent SERVAIS MD, PhD, Institut de Myologie, France
Other Study IDs: 2010-A00495-34
Record Dates: First submitted 2011-11-16; First posted 2011-11-18 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2011-11

CONDITIONS: Congenital Myasthenic Syndrome
Keywords: Congenital Myasthenic Syndrome; Pregnancy; Outcome
MeSH Terms: conditions — Myasthenic Syndromes, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a retrospective study that follows the clinical evolution, the pregnancy and the post-partum perioad of female patients with Congenital Myasthenic Syndrome.

DETAILED DESCRIPTION:
The aim of this study is to better understand the action of hormonal factors that are presumably incriminated for the fluctuation of the disease. The investigators would also like to better adress the issues of women with Congenital Myasthenic Syndrome, who desire a pregnancy : the possibility of decompensation, the problems that can arise during the course of the childbearing, the risk of foetal malformations.

ELIGIBILITY:
Inclusion criteria:

* Adult women
* Congenital myastenic syndrome genetically confirmed or with clinical compatible and electrophysiological evidence
* Written consent

Exclusion Criteria:

* Neurological or general pathology occurs significantly with the initiation and conduct of a pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with Congenital Myasthenie Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent SERVAIS, MD, PhD, Principal Investigator — institut myologie